CLINICAL TRIAL: NCT07214012
Title: Planning Together: A Couple-based, Multi-level Prenatal Contraceptive Education Program for Economically Marginalized Families
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Tennessee Graduate School of Medicine (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 5175; R21HD112736 (NIH)
Record Dates: First submitted 2025-10-01; First posted 2025-10-09 (Actual); Last update posted 2025-10-09 (Actual); Status verified 2025-10

CONDITIONS: Short Interpregnancy Intervals; Maternal Health Disparities

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Communication and Contraceptive Education Workbook (60-90 minutes) (Other): Asynchronous (during times convenient to the couple) (21-30 weeks gestation)
  Follow-up survey at the end of session
  Interventions: Other: Joint contraceptive and couple communication education
- Couple Contraceptive Consultation (60-90 minutes) (Other): In-person at OBGYN appt or telehealth (couple preference). ~ 32 weeks gestation
  Follow-up survey at the end of session
  Interventions: Other: Couple communication consultation with Interventionist to increase partner engagement and improve communication
- Booster Check-ins (~30 minutes) (Other): Telehealth/in-person (couple preference), ~6 weeks postpartum
  Follow-up survey at the end of sessions
  Interventions: Other: Check-ins to support continued partner support & communication
- Booster Check-ins (~30 minutes.) (Other): Telehealth/in-person (couple preference), ~12 weeks postpartum
  Follow-up surveys at the end of session
  Interventions: Other: Check-ins to support continued partner support & communication

INTERVENTIONS:
Other: Joint contraceptive and couple communication education — Joint Comprehensive Contraceptive Education
  a. Visual and written description of all currently available contraceptives with explanation of pros and cons
  Couple constructive communication education
  1. Specific couple contraceptive conversation examples.
  2. Interactive worksheet to help with joint desired contraceptive decision-making and making a consistent use plan
  Arms: Communication and Contraceptive Education Workbook (60-90 minutes)
Other: Couple communication consultation with Interventionist to increase partner engagement and improve communication — 1. Couples will bring their completed workbook to reference during the meeting and assess fidelity
  2. Reinforce couple contraceptive communication skills. Address any challenges couple has with skill implementation
  3. Review desired contraceptive method & consistent use plan
  4. Use motivational interviewing techniques to help couple agree on contraceptive plan
  Arms: Couple Contraceptive Consultation (60-90 minutes)
Other: Check-ins to support continued partner support & communication — 1. Review progress toward couple contraceptive communication skills and use of agreed contraceptive method
  2. Assess factors promoting successful contraceptive use and communication skills
  3. Address barriers to consistent contraceptive use and communication skill implementation via shared problem-solving
  Arms: Booster Check-ins (~30 minutes)
Other: Check-ins to support continued partner support & communication — 1. Review progress toward couple contraceptive communication skills and use of agreed contraceptive method
  2. Assess factors promoting successful contraceptive use and communication skills
  3. Address barriers to consistent contraceptive use and communication skill implementation via shared problem-solving
  Arms: Booster Check-ins (~30 minutes.)

SUMMARY:
The goal of this pilot trial is to examine the feasibility and acceptability of the Planning Together protocol

The hypothesis of this study are

1. The study will achieve feasibility, demonstrated by ≥80% study accrual (30 couples in 8 months), ≥75% protocol adherence, and ≥75% (e.g., education workbook completion)
2. The intervention will be acceptable, with >80% of participants reporting satisfaction with Planning Together.
3. Patterns of primary outcomes (contraceptive knowledge, communication quality, community referral utilization) and secondary outcomes (agreed contraceptive plan, consistent contraceptive usage and satisfaction, psychological distress, and Short Interpregnancy Intervals [SII]) will suggest benefits of the intervention.

DETAILED DESCRIPTION:
This study addresses critical maternal health disparities by targeting SII, which are associated with adverse outcomes such as preterm birth, low birth weight, and preeclampsia. These risks are especially high in economically marginalized populations, particularly in the Southern U.S., where access to prenatal contraceptive education is limited. The "Planning Together" intervention is a culturally-responsive, couple-based approach that seeks to improve consistent, desired contraceptive use by addressing both social barriers (e.g., lack of partner involvement and poor communication) and structural barriers (e.g., food insecurity, housing instability). It combines flexible delivery (online and in-person options) with tailored community referrals and partner-inclusive contraceptive education.

At approximately 20 weeks gestation, eligible pregnant participants will be recruited from the UT OBGYN Clinic, with their romantic partners recruited in-person or virtually. After informed consent, both participants will complete a baseline survey. This survey includes demographics and validated measures related to contraceptive knowledge, couple communication, reproductive autonomy, and psychological well-being. The visit also includes a social needs assessment using the Accountable Health Communities Screening Tool, which informs warm hand-off referrals during later sessions.

The significance of this work lies in its potential to reduce maternal health disparities through a brief (4-session), sustainable intervention model. If proven feasible and acceptable, "Planning Together" could be scaled to other underserved or marginalized communities and applied to additional perinatal health issues traditionally assigned to the pregnant-capable person (e.g., infant vaccinations, breastfeeding, peripartum mood disorders), ultimately improving both infant and maternal health outcomes.

ELIGIBILITY:
Inclusion Criteria:

Patient Inclusion Criteria:

1. > 20 weeks pregnant, age 18+
2. The pregnant person has an available romantic partner, and the couple was able to get pregnant on their own or will be able to after the delivery
3. separately, the pregnant person reports being in a sexually, psychologically and physically safe relationship
4. English-speaking

Romantic Partner Inclusion Criteria:

1. 18 years of age and older
2. Cohabiting with the patient; in a romantic relationship with patient
3. Capable of getting the patient pregnant after delivery
4. Does not need to be the biological father of the current pregnancy
5. English-speaking (in order to take part in the interview as the interviewer does not speak Spanish)

Exclusion Criteria:

Patient Exclusion Criteria:

1. Participant is under the age of 18
2. Documented cognitive impairment or psychiatric condition in pregnant person's medical record (e.g., severe learning disability, dementia, current psychotic disorder, suicidality)
3. Participation in a concurrent contraceptive education intervention
4. The pregnant person has a high-risk medical condition

Romantic Partner Exclusion Criteria:

1. Less than 18 years of age
2. Are not cohabiting with the patient; not in a romantic relationship with patient
3. Not capable of getting the patient pregnant after delivery

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-10-15 (Estimated); Primary Completion 2026-10-14 (Estimated); Study Completion 2026-10-14 (Estimated)

PRIMARY OUTCOMES:
Feasibility of Study Procedures | Baseline, 30 weeks gestation, 32 weeks gestation, 6-week postpartum, and 12-week postpartum
  Defined as ≥80% study accrual (30 couples in 8 months), ≥75% protocol adherence, and ≥75% fidelity (completion of workbook and study activities)
Acceptability of the Intervention | Baseline, 30 weeks gestation, 32 weeks gestation, 6-week postpartum, and 12-week postpartum
  Measured by survey item: >80% of participants will report satisfaction with Planning Together using a Program Satisfaction questionnaire
Change in Contraceptive Knowledge | Baseline, 30 weeks gestation, 32 weeks gestation, 6-week postpartum, and 12-week postpartum
  Measured using the validated Contraceptive Knowledge tool
Change in Couple Communication Quality | Baseline, 30 weeks gestation, 32 weeks gestation, 6-week postpartum, and 12-week postpartum
  Assessed with the Communication Problems Questionnaire (CPQ)
Community Referral Utilization | 32 weeks gestation to 12 weeks postpartum
  Community Referral Utilization and Satisfaction Questionnaire Scale (4 items validated by Dr. Roberson with economically marginalized couples

SECONDARY OUTCOMES:
Consistent Contraceptive Usage | 6-week postpartum and 12-week postpartum
  Measured by participant self-report on the Consistent Usage scale
Satisfaction with Agreed Contraceptive Method | 6-week postpartum and 12-week postpartum
  Assessed via the validated Satisfaction of Agreed Method scale
Relationship Satisfaction | Baseline, 30 weeks gestation, 32 weeks gestation, 6-week postpartum, and 12-week postpartum
  Measured using the Couple Satisfaction Index (CSI)
Psychological Distress - Anxiety | Baseline, 30 weeks gestation, 32 weeks gestation, 6-week postpartum, and 12-week postpartum
  Measured using PROMIS Anxiety short form
Psychological Distress - Depression | Baseline, 30 weeks gestation, 32 weeks gestation, 6-week postpartum, and 12-week postpartum
  Measured using PROMIS Depression short form
Relationship Aggression | Baseline, 30 weeks gestation, 32 weeks gestation, 6-week postpartum, and 12-week postpartum
  Measured using the Conflict Tactic Scale (CTS)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Tennessee Graduate School of Medicine, Knoxville, Tennessee, United States